CLINICAL TRIAL: NCT06128447
Title: A Phase 3, Multi-center, Prospective, Randomized, Double-blind, Placebo- Controlled Study to Evaluate the Effectiveness and Safety of ZP5-9676 for the Treatment of Hookworm (Ancylostoma Duodenale and Necator Americanus), Ascaris Lumbricoides, and Trichuris Trichiura in Pediatric and Adult Participants
Brief Title: Phase 3, Multi-center, Prospective, Randomized, Double-blind, Placebo- Controlled Study to Evaluate the Effectiveness and Safety of ZP5-9676 for the Treatment of Soil Transmitted Helminthiasis (STH)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zero Point Five Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZP5-9676-301
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Soil-Transmitted Helminthiasis (STH)

STUDY DESIGN:
Intervention Model Description: prospective, randomized, double-blind, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A (Active Comparator): ZP5-9676 600 mg dose
  Interventions: Drug: ZP5-9676 600 mg dose
- Treatment B (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ZP5-9676 600 mg dose — oral, chewable tablet formulation of flubendazole
  Arms: Treatment A
Drug: Placebo — Matching placebo
  Arms: Treatment B

SUMMARY:
This is a Phase 3, multi-center, prospective, randomized, double-blind, placebo-controlled study to evaluate the effectiveness, safety, and tolerability of ZP5-9676 compared to placebo for the treatment of STH infections. Approximately 300 participants will be enrolled, randomized at the Baseline visit (Day 1) to one of the following treatments in a 1:1 ratio of active and placebo.

DETAILED DESCRIPTION:
Approximately 300 infected participants will be enrolled to ensure that there is a minimum of 114 hookworm-infected participants evaluable for the Test of Cure study visit (Day 14). Some participants may be co-infected and will be included in each tally.

Participants will be randomized (1:1) to one of the treatments below followed by standard of care treatment:

* Treatment A: ZP5-9676 600 mg dose
* Treatment B: Placebo

ELIGIBILITY:
Inclusion Criteria:

1. Provide a signed informed consent form from the participant or parent/guardian, and assent by participant(as applicable per local requirements) and understand and agree to comply with required procedures in the study.
2. Male or female, who are 6 months to 59 years old, inclusive, and live in a high STH prevalence area
3. Positive for hookworm (A. duodenale or N. americanus), A. lumbricoides, and/or T. trichiura on microscopic examination of fecal samples.
4. Females of childbearing potential must use an acceptable method of contraception as determined by the Investigator from the initial Screening visit through 35 days after study drug administration. A female is considered to be of childbearing potential from menarche until after menopause (age >45 years with no menses for 12 months without an alternative medical cause) unless permanently sterile. Acceptable methods include abstinence, hormonal contraceptives, intrauterine device/system, vasectomy in the sole male sexual partner, tubal ligation, or double-barrier contraceptive method (male condom with female cervical cap, diaphragm, or sponge) with spermicide.
5. Otherwise healthy based on medical history, physical examination, vital signs, and concomitant medications for inclusion.

Exclusion Criteria:

1. Severe anemia (hemoglobin< 8 g/dL1).
2. Active diarrhea (passage of ≥3 loose or liquid stools per day).
3. Children (6 months to 17 years old) with significant wasting (moderate and severe-below minus two standard deviations from median weight for height of reference population).
4. Women who are pregnant.
5. Hypersensitivity or allergy to ZP5-9676 or any inert ingredients in the chewable formulation or other medications in the benzimidazole class.
6. Taken ZP5-9676 or any other treatment for STH infection within 30 days of screening or randomization.
7. Used an investigational medical device within 30 days of screening.
8. Preplanned surgery procedures within 30 days of screening.
9. History of a medical disorder causing difficulty in chewing or swallowing.
10. Participation in any investigational drug (including vaccine) trial within 30 days or six half-lives of the test drug's biologic activity, whichever is longer, before the start of the study (time of first dose).
11. Participation in an interventional clinical study within 30 days of screening.
12. Any condition that interferes with the ability to understand or comply with the requirements of the study.
13. Any other medical condition, serious illness, or other circumstance that would place the subject at increased risk, as determined by the Investigator

Ages: 6 Months to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cure rates | 14 days
  Cure rates (CRs) for each STH

SECONDARY OUTCOMES:
Egg reduction | 14 days
  Egg reduction rates (ERRs) for hookworm
Cure rates | 14 days
  Cure rates of hookworm

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica de Vacinas, Americaninha, Brazil

IPD SHARING:
Plan to Share IPD: No